CLINICAL TRIAL: NCT03533049
Title: mHealth Family Self-Management Intervention for Parents of Transplanted Children
Brief Title: mHealth Family Self-Management
Acronym: myFAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Stacee Lerret, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 1183697
Record Dates: First submitted 2018-04-25; First posted 2018-05-22 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Transplantation; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myFAMI intervention (Experimental): All participants will receive the standard discharge education from their transplant and inpatient care team.
  Patients who are assigned to the myFAMI group will also have the smartphone application downloaded onto either the family member's smartphone or a study-provided smartphone. Following discharge from the hospital, participants will use the smartphone application to answer nine daily questions regarding tracking family coping, transplant symptoms, family management of child transplant symptoms, and family-management difficulty with medication and follow-up regimen daily for the first 30 days following discharge.
  Interventions: Other: myFAMI
- Control (Active Comparator): Family members assigned to the control group (standard care) will receive standard post-discharge follow-up care consisting of discharge education during the transplant hospitalization and at regularly scheduled appointments instructing families to contact the research nurse with problems or questions.
  Interventions: Other: myFAMI

INTERVENTIONS:
Other: myFAMI — Patients who are assigned to the myFAMI group will also have the smartphone application downloaded onto either the family member's smartphone or a study-provided smartphone. Following discharge from the hospital, participants will use the smartphone application to answer nine daily questions regarding tracking family coping, transplant symptoms, family management of child transplant symptoms, and family-management difficulty with medication and follow-up regimen daily for the first 30 days following discharge.

SUMMARY:
This innovative research will address a gap in the literature involving the evaluation of the impact of an individualized family-centered mHealth application to enhance daily post-discharge communication following pediatric transplant. This proposal lays the foundation for future research with myFAMI (self-management intervention) at multiple pediatric transplant centers and builds the science from which to consider post discharge monitoring and decrease cost of care in other pediatric chronic illness populations.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients:

1. Has undergone a heart, kidney, or liver transplant being discharged home from the hospital
2. Has two eligible family members available to answer questions about the patient

Family members will be eligible for participation upon meeting the following inclusion criteria:

1. is English speaking (to date the instruments being used have been validated for English speaking participants only)
2. is 18 years of age or older
3. has a pediatric family member (< 18 years old) who has undergone a heart, kidney, or liver transplant being discharged home from the hospital.

Exclusion Criteria for the family members are:

1. presence of significant communication or cognitive impairment that would preclude completion of questionnaires based on self-report; or
2. the pediatric family member has experienced a previous transplant based on self report.

Participants unable to speak and read English will be excluded due to the lack of resources to develop the app and communicate via FaceTime in different languages. We will recruit family members from three types of transplant populations to allow for sufficient sample in a limited time frame for this complex pediatric surgery and high-risk population.

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Improve family coping | 30 days
  Primary family member receiving myFAMI compared to the primary family member receiving standard post-discharge care will have improved post-discharge coping (primary outcome). Coping will be measured using the post-discharge coping difficulty scale. Post Discharge Coping Difficulty Scale (PDCDS), 10-item measure, Scale 0-10, Measures parental and family member difficulty coping with stress, recovery, self-care and management, support, and confidence, α= .84

SECONDARY OUTCOMES:
Decrease healthcare resources | 30 days
  Primary family member receiving myFAMI compared to the primary family member receiving standard post-discharge care will have decreased use of healthcare resources defined as number of emergency department visits and number or readmissions to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lerret SM, Flynn E, White-Traut R, Alonso E, Mavis AM, Jensen MK, Peterson CG, Schiffman R. Acceptability of an mHealth Family Self-management Intervention (myFAMI) for Pediatric Transplantation Families: Qualitative Focus. JMIR Nurs. 2022 Jul 15;5(1):e39263. doi: 10.2196/39263. PMID 35838761